CLINICAL TRIAL: NCT06241794
Title: Comparison of Postoperative Analgesic Efficacy of Perichondrial Approach Modified Thoracoabdominal Nerve Block and the Combination of Serratus Intercostal Plane and Rectus Sheath Block Via to Patients Who Underwent Cholecystectomy
Brief Title: The Efficacy of Thoracoabdominal Nerve Block With Serratus Intercostal Plane and Rectus Sheath Block in Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Güvenç Doğan, associated professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-172
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pain Management
Keywords: Laparoscopic Cholecystectomy; Modified Thoracoabdominal Plane Block; Serratus Intercostal Plane Block; Rectus Sheath Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Active Comparator): M-TAPA:
  Aseptic conditions are ensured in the area where the block will be performed. Under ultrasound guidance, a linear probe at the sagittal plane and costochondral angle is used to identify the transversus abdominis, internal oblique, and external oblique muscles at the level of the 10th rib. To visualize the lower surface of the rib cartilage in the midline, a sagittal angle is applied with the probe in the direction of the costochondral angle at the edge of the 10th rib. Using a 22-G, 80-100 mm block needle with an in-plane technique, the needle is advanced cranially. The needle tip is directed towards the posterior surface of the 10th rib cartilage, underneath the condyle. Subsequently, 20 ml of 0.25% concentration bupivacaine is injected beneath the condyle. The same procedure will be applied to the opposite side using the same technique.
  Interventions: Procedure: Group M-TAPA
- Group Serratus Intercostal Plane Block and Rectus Sheath Block (Active Comparator): Serratus intercostal plane block:The serratus anterior muscle and intercostal muscles are identified at the level of 8th rib along the right mid-axillary line.Using block needle,20 ml of 0.25% Bupivacaine is injected into the interfascial plane between these muscles.The SIPB will be performed only on right side.
  Rectus sheath block:a linear probe is placed in a transverse position just above the umbilicus and slightly lateral to the midline.After visualizing the rectus abdominis muscle, posterior rectus sheath,and the hypoechoic space between them,block needle is advanced in-plane along the subcutaneous tissue.The needle is progressed until reaching the space between the epimysium of the muscle and the posterior rectus sheath, passing horizontally through the anterior rectus sheath of the rectus abdominis muscle.10 ml of 0.25% bupivacaine is injected.Adequate spread will lift the epimysium of the rectus abdominis muscle while displacing the posterior fascia and peritoneum downward
  Interventions: Procedure: Group Serratus Intercostal Plane Block and Rectus Sheath Block

INTERVENTIONS:
Procedure: Group M-TAPA — Aseptic conditions are ensured in the area where the block will be performed. Under ultrasound guidance, a linear probe at the sagittal plane and costochondral angle is used to identify the transversus abdominis, internal oblique, and external oblique muscles at the level of the 10th rib. To visualize the lower surface of the rib cartilage in the midline, a sagittal angle is applied with the probe in the direction of the costochondral angle at the edge of the 10th rib. Using a 22-G, 80-100 mm block needle with an in-plane technique, the needle is advanced cranially. The needle tip is directed towards the posterior surface of the 10th rib cartilage, underneath the condyle. Subsequently, 20 ml of 0.25% concentration bupivacaine is injected beneath the condyle. The same procedure will be applied to the opposite side using the same technique.
  Arms: Group M-TAPA
Procedure: Group Serratus Intercostal Plane Block and Rectus Sheath Block — Serratus intercostal plane block:The serratus anterior muscle and intercostal muscles are identified at the level of 8th rib along the right mid-axillary line.Using block needle,20 ml of 0.25% Bupivacaine is injected into the interfascial plane between these muscles.The SIPB will be performed only on the right side.
  Rectus sheath block:a linear probe is placed in a transverse position just above the umbilicus and slightly lateral to the midline.After visualizing the rectus abdominis muscle, posterior rectus sheath,and the hypoechoic space between them,block needle is advanced in-plane along the subcutaneous tissue.The needle is progressed until reaching the space between the epimysium of the muscle and the posterior rectus sheath, passing horizontally through the anterior rectus sheath of the rectus abdominis muscle.10 ml of 0.25% bupivacaine is injected.Adequate spread will lift the epimysium of rectus abdominis muscle while displacing the posterior fascia and peritoneum downward
  Arms: Group Serratus Intercostal Plane Block and Rectus Sheath Block

SUMMARY:
Cholecystectomy is a widespread surgical procedure performed worldwide for acute cholecystitis. This operation can be performed using open surgery or laparoscopic techniques. Laparoscopic technique is superior to open surgery in terms of less pain at incision sites, shorter hospital stay, improved quality of life, and faster recovery times.However, despite being a minimally invasive surgery, laparoscopic cholecystectomy (LC) can still cause moderate to severe pain. Severe pain can lead to delayed postoperative ambulation, decreased patient satisfaction, the development of chronic pain, and is associated with increased lung and heart complications. Postoperative pain in LC can stem from various causes. To reduce the postoperative pain caused by LC, non-steroidal anti-inflammatory drugs, paracetamol, opioids, local anesthetics, and various regional anesthesia techniques are used.Multimodal analgesia has shown that the use of regional anesthesia and analgesia is crucial in reducing the neuroendocrine stress response in pain and trauma situations. The use of interfascial plane blocks performed under ultrasound guidance in LC surgery, considered easy and safe, has increased in recent years. The thoracoabdominal plane block (TAPA) applied through a perichondrial approach reaches a broader dermatomal area than the transversus abdominis plane (TAP) block and the oblique subcostal transversus abdominis plane (OSTAP) block.Serratus intercostal plane block (SIPB) has been found effective for somatic analgesia in a case series after gastrectomy and cholecystectomy surgeries. Subsequent studies have indicated the effectiveness of SIPB for open upper abdominal surgeries. Rectus sheath block (RSB) is used to provide postoperative analgesia after various surgeries, including laparoscopic and upper abdominal surgeries. Ultrasound-guided RSB in LC has significantly reduced postoperative pain.In this study, similar to the combination of RSB and SIPB was planned to be applied to enhance the effectiveness and quality of analgesia in the mid-abdomen. A group in LC surgery was administered bilateral M-TAPA, while another group received bilateral RSB + right SIPB, aiming to compare the postoperative analgesic effectiveness.

DETAILED DESCRIPTION:
The gallbladder is a small organ located in the right upper quadrant of the abdomen. Bile, which aids in the digestion of food, is collected in this organ. Gallstones are solid particles that form as a result of changes in the composition and concentration of bile caused by hormones, medications, diet, and weight changes. Sometimes, gallstones that form can block the normal flow of bile by exiting the gallbladder, leading to a condition known as acute cholecystitis when the cystic duct is obstructed by a gallstone. This condition causes distension and inflammation of the gallbladder.

Cholecystectomy is a common surgical procedure performed worldwide for acute cholecystitis. The management of acute cholecystitis is divided into medical and surgical approaches. Medical management includes bed rest, analgesic agents, antibiotic therapy, and intravenous fluid replacement. Surgical management involves a procedure called cholecystectomy, which is the surgical removal of the gallbladder. This operation can be performed using open surgery or laparoscopic techniques. The laparoscopic technique is superior to open surgery in terms of less pain at incision sites, shorter hospital stay, improved quality of life, and faster recovery times. However, laparoscopic cholecystectomy (LC), despite being a minimally invasive surgery, can still cause moderate to severe pain.

Severe pain can lead to delayed postoperative ambulation, decreased patient satisfaction, the development of chronic pain, and is associated with increased lung and heart complications. Postoperative pain in LC can arise from various causes. While a significant portion of postoperative pain in LC is attributed to incision sites (50-70%), it also originates from pneumoperitoneum (20-30%) and cholecystectomy (10-20%). Multimodal analgesia, including non-steroidal anti-inflammatory drugs, paracetamol, opioids, local anesthetics, and various regional anesthesia techniques, should be considered for pain control. Opioids may cause side effects such as postoperative nausea and vomiting (PONV), constipation, and respiratory depression. Neuraxial analgesia is rarely used in LC due to possible complications and technical difficulties.

The use of interfascial plane blocks under ultrasound guidance, considered easy and safe, has increased in LC surgery. The thoracoabdominal plane block (TAPA) applied through a perichondrial approach, showing that it spreads to a broader dermatomal area than the transversus abdominis plane (TAP) block and the oblique subcostal transversus abdominis plane (OSTAP) block. The rectus sheath block (RSB) is used to provide postoperative analgesia after various surgeries, including laparoscopic and upper abdominal surgeries. Ultrasound-guided RSB in LC has significantly reduced postoperative pain.

In this study, the combination of RSB and SIPB was planned to be applied to enhance the effectiveness and quality of analgesia in the mid-abdomen. Patients will be asked to fill out the Quality of Recovery-15 (QoR-15) scale, a self-report questionnaire used to assess the quality of postoperative recovery, in the preoperative waiting area on the morning of the surgery and 24 hours after the surgery. The QoR-15 scale measures recovery quality in five areas: physical comfort, pain, physical independence, psychological support, and emotional state, providing a one-dimensional measurement of recovery quality with scores ranging from 0 to 150. A higher score indicates better recovery quality.

In this study, in laparoscopic cholecystectomy, one group will receive bilateral M-TAPA, and another group will receive bilateral RSB + right SIPB to investigate their superiority in terms of postoperative NRS (Numeric Rating Scale) score, opioid consumption, dermatomal spread, PONV score, and complications, aiming to determine which is more effective.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification with physical status 1-2
* Between the ages of 18 and 65
* Body Mass Index (BMI) <35
* Has read and accepted the informed consent form voluntarily

Exclusion Criteria:

* The patient's unwillingness to participate in the study
* Patients with a body mass index (BMI) >35
* ASA 3-5 classification
* unable to use the NRS pain scoring system
* allergies to the used local anesthetic and specified analgesic drugs
* individuals declaring pregnancy or breastfeeding
* patients under 18 or over 65 years of age
* those with uncontrolled anxiety
* alcohol and drug addiction
* neuromuscular and peripheral nerve diseases
* using high-dose opioid drugs three days before surgery
* hepatic and renal insufficiency, coagulation disorders
* diabetes mellitus
* patients using anticoagulant drugs
* infections at the site of peripheral block needle entry
* those undergoing a second procedure along with laparoscopic cholecystectomy
* individuals with a history of abdominal surgery or trauma
* conversion of laparoscopic surgery to open surgery
* inability to communicate in Turkish
* NRS score above 7 for consecutive 4 hours despite the planned multimodal analgesia regimen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-08-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group M-TAPA: M-TAPA:
  Group M-TAPA: Aseptic conditions are ensured in the area where the block will be performed. Under ultrasound guidance, a linear probe at the sagittal plane and costochondral angle is used to identify the transversus abdominis, internal oblique, and external oblique muscles at the level of the 10th rib. To visualize the lower surface of the rib cartilage in the midline, a sagittal angle is applied with the probe in the direction of the costochondral angle at the edge of the 10th rib. Using a 22-G, 80-100 mm block needle with an in-plane technique, the needle is advanced cranially. The needle tip is directed towards the posterior surface of the 10th rib cartilage, underneath the condyle. Subsequently, 20 ml of 0.25% concentration bupivacaine is injected beneath the condyle. The same procedure will be applied to the opposite side using the same technique.
Period: Overall Study
Arm/Group | Group M-TAPA | Group Serratus Intercostal Plane Block and Rectus Sheath Block
Started | 35 | 37
Completed | 35 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group M-TAPA | Group Serratus Intercostal Plane Block and Rectus Sheath Block | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 0 | 0 | 0
Age, Continuous [Geometric Least Squares Mean (Inter-Quartile Range); unit: year] | 44 [19 to 68] | 45 [19 to 68] | 45 [19 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Examination
Description: Determination of patients' post-operative pain level. The Numeric Rating Scale (NRS), a method that converts the patient's pain perception into a numerical form, will be used to assess postoperative pain. NRS has a numerical scale ranging from 0 to 10. The patient will rate the intensity of pain on a scale from 0, indicating no pain, to 10, representing the worst imaginable pain (NRS 0=no pain, 4=mild to moderate pain, 6-8=severe pain, and >8=intolerable pain). The NRS score will be evaluated both at rest and during active movement situations (such as transitioning from a lying to a sitting position).
  The Numeric Rating Scale (NRS): (NRS 0=no pain, 4=mild to moderate pain, 6-8=severe pain, and >8=intolerable pain)
Time Frame: 24 hour
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Group M-TAPA | Group Serratus Intercostal Plane Block and Rectus Sheath Block
Number analyzed (Participants) | 35 | 37
score on a scale
  0th hour Rest NRS | 3 [1 to 6] | 5 [0 to 8]
  1th hour Rest NRS | 2 [0 to 4] | 3 [0 to 6]
  3th hour Rest NRS | 2 [0 to 5] | 2 [1 to 4]
  6th hour Rest NRS | 1 [0 to 3] | 2 [0 to 5]
  12th hour Rest NRS | 1 [0 to 3] | 2 [0 to 4]
  18th hour Rest NRS | 1 [0 to 3] | 1 [0 to 5]
  24th hour Rest NRS | 1 [0 to 3] | 2 [0 to 4]
  0th hour Active NRS | 4 [2 to 8] | 6 [1 to 9]
  1th hour Active NRS | 3 [1 to 6] | 4 [2 to 6]
  3th hour Active NRS | 3 [1 to 6] | 3 [1 to 6]
  6th hour Active NRS | 2 [1 to 4] | 3 [1 to 6]
  12th hour Active NRS | 2 [1 to 4] | 3 [1 to 4]
  18th hour Active NRS | 2 [0 to 4] | 2 [1 to 6]
  24th hour Active NRS | 2 [0 to 3] | 3 [1 to 4]

2. Secondary Outcome: Opioid Consumption
Description: Total 24-hour tramadol consumption of patients in mg.
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Group M-TAPA | Group Serratus Intercostal Plane Block and Rectus Sheath Block
Number analyzed (Participants) | 35 | 37
mg | 92.64 (26.28) | 103.9 (39.32)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Group M-TAPA | Group Serratus Intercostal Plane Block and Rectus Sheath Block
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 6/35 | 7/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group M-TAPA (N=35) | Group Serratus Intercostal Plane Block and Rectus Sheath Block (N=37)
Nausea or Vomiting (Gastrointestinal disorders) | 6 | 7 — Patients were followed up with the postoperative nausea and vomiting (PONV) scale in the first 24 hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT06241794/Prot_SAP_000.pdf